CLINICAL TRIAL: NCT03610503
Title: The Effect of Preferred Music on Anxiety and Pain in Electrodiagnostic Studies: A Prospective Randomized Trial
Brief Title: The Effect of Preferred Music on EMG Anxiety and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REDA 5189
Record Dates: First submitted 2018-07-12; First posted 2018-08-01 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Anxiety; Pain; Nerve Injury
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, intervention-control, trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Anonymous data collection to be reviewed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Patients listen to music during EMG test
  Interventions: Other: Music
- Control (Standard Care) (No Intervention): Patients do not listen to music during EMG test (ie. Standard of care)

INTERVENTIONS:
Other: Music — Participants in this arm will listen to music during the EMG testing
  Arms: Music

SUMMARY:
Patients often report anxiety and pain related to electromyography (EMG) and nerve conduction studies (NCS) which are tests used to look for diseases of the nerves and muscles. Unfortunately, for those with very high levels of test related stress, the experience may be very frightening and may impede completion of the study and negatively impact on making a timely and accurate diagnosis. Several studies have shown that music can improve anxiety and pain levels in various situations and procedures. Our study will allow participants to play music of their choice during EMG and NCS in order to determine if the pain and anxiety that they experience is reduced.

DETAILED DESCRIPTION:
This study will be a prospective randomized trial carried out at Mount Hope Centre for Long Term Care in London, Ontario. All patients referred for electromyography and a nerve conduction study will be considered for inclusion in the study. Those who meet the criteria and verbally consent to the study will sign a consent form and then be randomly assigned to either a music or no-music group using a computer-generated random number series. Prior to starting the test, all participants who enroll in the study will complete form Y-1 and Y-2 of the state-trait anxiety inventory (STAI) which measure state (S) anxiety and trait (T) anxiety respectively. They will also complete an 100 mm visual analogue scale (VAS) for pain and anxiety prior to beginning the studies. During and following the test they will be asked to complete a VAS for pain and anxiety, and the Y-1 of the STAI to measure state anxiety. Aside from having to fill out the STAI and visual analogue scales, patients assigned to the no-music group will undergo the EMG and NCS as per usual. Those in the music group will be given a set of over-ear headphones (sterilized before use) and a tablet device. Participants will be allowed to navigate Spotify, a digital music service to select whatever music they desire. An app that limits volume will be used to ensure that volume cannot be raised above 80 decibels by the patient. Communication with the patient will not be hindered as the EMG technician and physician will be speaking into a microphone that transmits the sound directly to the participant's headphones.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older referred for NCS and EMG at Mount Hope Centre for Long Term Care in London, Ontario will be eligible and offered entry into the study if the following criteria are met: the NCS/EMG are indicated, they have at least a 6th grade reading level in English such that they can complete the STAI, and the patient is willing and able to provide signed informed consent.

Exclusion Criteria:

1. Use of hearing aids that would preclude or hinder the use of over-ear headphones.
2. Profound hearing loss.
3. Cognitive Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
State-trait anxiety inventory (STAI) | Change in STAI (State sub-scale) from immediately before the EMG procedure, during the EMG procedure and immediately after EMG procedure
  Anxiety inventory that measures both Trait (T) and State (S) anxiety. Each sub- scale (T and S) is measured from 20-80 and reported individually (not combined) with higher values indicating higher anxiety. The typical cut off for S sub-scale is a score greater than 40 indicating clinically significant symptoms.

SECONDARY OUTCOMES:
Visual analog scale (VAS) for pain and anxiety scale (0-100) | Change in VAS immediately before the EMG procedure, during the EMG procedure, and immediately after EMG procedure
  Pain and anxiety scale using a standard VAS (0 = No pain/anxiety, 100 = maximal).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Macaluso, M.D., Principal Investigator — Schulich School of Medicine and Dentistry
Locations (1):
- Mount Hope EMG Lab, St. Joseph's Health Care (SJHC), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No